CLINICAL TRIAL: NCT06003127
Title: REcovery From DEXmedetomidine-induced Unconsciousness
Acronym: REDEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Emery Brown, Professor of Anesthesia, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P001821
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Healthy; Consciousness, Level Altered
Keywords: Dexmedetomidine; EEG; Transcranial magnetic stimulation; Cognition
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS-EEG Arm (Experimental): This arm will undergo TMS-EEG during the study.
  Interventions: Device: Transcranial Magnetic Stimulation-Electroencephalography
- Non-TMS-EEG Arm (No Intervention): This arm will not undergo TMS-EEG during the study.

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation-Electroencephalography — Transcranial magnetic stimulation of the cerebral cortex and measurement of TMS-evoked potentials in the EEG.
  Other Names: TMS-EEG
  Arms: TMS-EEG Arm

SUMMARY:
This pilot study in healthy volunteers aims to determine if biological sex has an impact on recovery from dexmedetomidine-induced unconsciousness, and if transcranial magnetic stimulation combined with electroencephalography (TMS-EEG) can be used to measure brain complexity during dexmedetomidine sedation without arousing study participants.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 65
* Normal body weight and habitus, body mass index (BMI) 18 to 30 kg/m2
* Non-smoker
* No history of taking stimulants or substance abuse
* For women: either use of hormonal contraception, or > 45 years old and last menstrual period > 12 months ago in the absence of any contraceptives.
* American Society of Anesthesiologists (ASA) physical status classification 1 (ASA 1)
* Fluent in English (sufficient to communicate with the study team and understand the consent form)

Exclusion Criteria:

* Neurologic: epilepsy or positive history of a seizure, stroke, central disorders of hypersomnolence, neuroimmunological disorder (e.g. multiple sclerosis), Meniere's disease, Parkinson's disease, peripheral neuropathy, no significant visual or hearing impairments, findings in the clinical examination suggesting a neurologic disorder
* Psychiatric: history or treatment for an active psychiatric problem (including Attention-Deficit / Hyperactivity Disorder (ADHD) and anxiety disorder)
* Cardiovascular: hypertension, symptomatic hypotension or bradycardia, myocardial infarction, coronary artery disease, peripheral vascular disease, dysrhythmias, congestive heart failure, cardiomyopathy, valvular disease, familial history of sudden cardiac death
* Respiratory: bronchitis, asthma, chronic obstructive pulmonary disease, smoking, shortness of breath, sleep apnea
* Gastrointestinal: esophageal reflux, hiatal hernia, ulcer
* Hepatic: hepatitis, jaundice, ascites
* Renal: acute or chronic severe renal insufficiency
* Reproductive: pregnancy, breast-feeding
* Endocrine: diabetes, thyroid disease, adrenal gland disease
* Hematologic: blood dyscrasias, anemia, coagulopathies
* Musculoskeletal: prior surgery or trauma to head neck or face, arthritis, personal or family history of malignant hyperthermia
* Medications: regular use of prescription and non-prescription medications expected to affect central nervous function, anticoagulant or thrombocyte-aggregation inhibiting therapy; exception: oral hormonal contraception
* Allergies: dexmedetomidine, phenylephrine, betablockers (including labetalol and esmolol), hydralazine, glycopyrrolate

Potential participants will not be enrolled in our study if they fail to pass a standard drug screening test (toxicology).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to return of responsiveness | Up to 120 minutes
  The time to return of responsiveness will be measured in minutes and from the moment of dexmedetomidine discontinuation to the return of clicking a button in response to auditory stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Emery N Brown, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vincent KF, Mallari OG, Dillon EJ, Stewart VG, Cho AJ, Dong Y, Edlow AG, Ichinose F, Xie Z, Solt K. Oestrous cycle affects emergence from anaesthesia with dexmedetomidine, but not propofol, isoflurane, or sevoflurane, in female rats. Br J Anaesth. 2023 Jul;131(1):67-78. doi: 10.1016/j.bja.2023.03.025. Epub 2023 May 2. PMID 37142466
- [Background] Kato R, Zhang ER, Mallari OG, Moody OA, Vincent KF, Melonakos ED, Siegmann MJ, Nehs CJ, Houle TT, Akeju O, Solt K. D-Amphetamine Rapidly Reverses Dexmedetomidine-Induced Unconsciousness in Rats. Front Pharmacol. 2021 May 18;12:668285. doi: 10.3389/fphar.2021.668285. eCollection 2021. PMID 34084141